CLINICAL TRIAL: NCT03348566
Title: Fish and Marine Fatty Acids, Genetic Signatures of Diet Adaptation, and Long-term Weight Change
Brief Title: Fish and Marine Fatty Acids, Genetic Signatures of Diet Adaptation, and Long-term Weight Changes
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Other Study IDs: NHS25487541
Record Dates: First submitted 2017-10-26; First posted 2017-11-21 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — In Situ Hybridization, Fluorescence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: fish — fish intkae

SUMMARY:
the investigators tested whether genetic variants near FADS cluster, which were recently identified to be signatures of adaptation to fish- and n-3 PUFAs-rich diet, interacted with these dietary factors on long-term change of body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* 11,323 women of European ancestry.
* Informed consent was obtained from all participants. The DNA extraction methods, quality control measures,
* SNPs genotyping and imputation data are available .
* Both cases and controls with genotyping data are available based on GWASs

Exclusion Criteria:

* participants without genetic data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Nurses' Health Study began in 1976, when 121,700 female registered nurses aged 30-55 y were recruited to complete a baseline questionnaire. the investigators included 11,323 women of European ancestry. Informed consent was obtained from all participants.
  The Health Professionals Follow-up Study The HPFS was initiated in 1986, and was composed of 51,529 male aged 40-75 y at baseline. This study included 6,833 men whose genotype data were available. Informed consent was obtained from all participants.
  The Women's Health Initiative (WHI) is a large, multiethnic, 40-center study that focuses on strategies for preventing heart disease, breast and colorectal cancer, and osteoporotic fractures in postmenopausal women. 6,254 Caucasians women with European ancestry were included.
  The design of Singapore Chinese Health Study (SCHS): Between 1993 and 1998, 63,257 Chinese between 45 and 74 in Singapore were enrolled. 5,264 subjects with genotyping data were included in this analysis.
Sampling Method: Non-Probability Sample
Enrollment: 22000 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
weight changes | 6-10 years
  long term weight changes: this study measured body weight at baseline (1990) and follow up body weight in 2000. The long term body weight was defined as changes from baseline to follow up endpoint

IPD SHARING:
Plan to Share IPD: No
The data belongs to HSPH

REFERENCES:
- [Background] Heianza Y, Qi L. Gene-Diet Interaction and Precision Nutrition in Obesity. Int J Mol Sci. 2017 Apr 7;18(4):787. doi: 10.3390/ijms18040787. PMID 28387720
- [Background] Qi Q, Chu AY, Kang JH, Huang J, Rose LM, Jensen MK, Liang L, Curhan GC, Pasquale LR, Wiggs JL, De Vivo I, Chan AT, Choi HK, Tamimi RM, Ridker PM, Hunter DJ, Willett WC, Rimm EB, Chasman DI, Hu FB, Qi L. Fried food consumption, genetic risk, and body mass index: gene-diet interaction analysis in three US cohort studies. BMJ. 2014 Mar 19;348:g1610. doi: 10.1136/bmj.g1610. PMID 24646652